CLINICAL TRIAL: NCT01932476
Title: Randomized Double-Masked Gluten Challenge to Evaluate Markers of Autoimmunity in Patients With Type-1 Diabetes and Celiac Disease After Oral Gluten Challenge
Brief Title: Gluten Immunity and Islet Autoimmunity in Type-1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: ImmusanT, Inc. (Industry)
Responsible Party: Principal Investigator, Jason Gaglia, Assistant Investigator, Joslin Diabetes Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: GC001
Record Dates: First submitted 2013-08-14; First posted 2013-08-30 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes; Celiac Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Celiac Disease Alone Gluten Challenge (Experimental)
  Interventions: Dietary Supplement: Gluten Challenge
- Celiac Disease Alone Sham Challenge (Sham Comparator)
  Interventions: Dietary Supplement: Sham Challenge
- Celiac Disease and T1D Gluten Challenge (Experimental)
  Interventions: Dietary Supplement: Gluten Challenge
- Celiac Disease and T1D Sham Challenge (Sham Comparator)
  Interventions: Dietary Supplement: Sham Challenge

INTERVENTIONS:
Dietary Supplement: Gluten Challenge — Three-day gluten containing dietary challenge.
  Arms: Celiac Disease Alone Gluten Challenge; Celiac Disease and T1D Gluten Challenge
Dietary Supplement: Sham Challenge — Three-day sham (gluten free) dietary challenge
  Arms: Celiac Disease Alone Sham Challenge; Celiac Disease and T1D Sham Challenge

SUMMARY:
The purpose of this study is to determine whether the immune response causing celiac disease is related to the autoimmune response causing type-1 diabetes.

DETAILED DESCRIPTION:
Participants meeting eligibility criteria will have blood collected before and after a three-day oral gluten challenge. This blood will be tested for biomarkers associated with islet autoimmunity and gluten-specific cellular immunity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Celiac Disease by histology and serology
* For those with Type-1 Diabetes, at least one anti-islet antibody
* HLA-DQ2.5 genotype

Exclusion Criteria:

* Not following a gluten free diet for at least 12 months
* Known gluten exposure within the prior 2 months
* Treatment with systemic immune modifying biological agents (adalimumab, etanercept, infliximab, certolizumab pegol) in prior 6 months
* Treatment with systemic immunomodulatory agents in prior 30 days
* Human immunodeficiency virus infection, untreated hepatitis B virus, or hepatitis C virus infection
* Nut allergy
* Hemoglobin level below normal range
* History of angina
* Pregnant or lactating
* Severe symptoms to gluten challenge in the past
* Elevation in transglutaminase-IgA or deamidated gliadin peptide IgA or IgG greater than or equal to 50% above upper limit of normal
* Uncontrolled complications of type-1 diabetes or celiac disease which pose a risk to participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Markers of Autoimmunity | Baseline and day 3 post challenge
  Blood samples for markers of autoimmunity will be taken before and day 3 post challenge.

SECONDARY OUTCOMES:
Gastrointestinal Symptoms | Baseline and 6 days
  Gastrointestinal symptoms are recorded in a standardized diary at baseline and for 6 days inclusive of challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gaglia, MD, MMSc, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States